CLINICAL TRIAL: NCT03575312
Title: Pharmacokinetic Study to Assess and Compare the Pharmacokinetics of Enrofloxacin After Dermal, Inhaled, and Oral Dosing
Brief Title: Pharmacokinetics of Enrofloxacin in Plasma and Urine
Acronym: EnroHuman
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Collaborators: Federal Institute for Occupational Safety and Health (BAuA)/Germany) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18-02 EnroHuman
Record Dates: First submitted 2018-05-30; First posted 2018-07-02 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Healthy
MeSH Terms: interventions — Enrofloxacin

STUDY DESIGN:
Intervention Model Description: The subjects are exposed to 250 µg of enrofloxacin on three different dosing days that are separated by at least 7 days. On the first dosing day, enrofloxacin is administered via the dermal route. On the second dosing day, enrofloxacin is administered via inhalation of 5 mL solution in a concentration of 50 µg/mL by an ultrasonic nebulizer. On the third dosing day, enrofloxacin is administered orally as a 20 mL solution in a concentration of 12.5 µg/mL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enrofloxacin (Experimental): enrofloxacin by dermal route, by inhalation, oral adminstration
  Interventions: Drug: Enrofloxacin

INTERVENTIONS:
Drug: Enrofloxacin — dermal application, inhalation rsp. oral administration of Enrofloxacin

SUMMARY:
Antibiotics like enrofloxacin are widely used in animal farming to treat and prevent bacterial infections. A previous study in poultry farms has shown that yardmen show significant concentrations of administered antibiotics in their urine. It is currently unclear how poultry yardmen are exposed to the administered antibiotics. The objective of this exemplarily study is to obtain information on the pharmacokinetics of the different uptake routes (oral, inhaled or dermal).

DETAILED DESCRIPTION:
Study subjects will be exposed to enrofloxacin at a concentration level representative for occupational exposure of yardmen at poultry farms.

As three uptake-routes, oral, inhalation and dermal, are conceivable all three cases will be investigated. After administration blood and urine samples will be analysed for enrofloxacin and its main metabolite ciprofloxacin at several time points. The objective of this exemplarily study is to obtain information on the pharmacokinetics of the different uptake routes. If different exposure routes are characterized by different pharmacokinetics, such studies can be used to obtain a better understanding of general routes of exposure in occupational environments. On the basis of the results mitigation strategies can be developed, reducing the risk of exposure.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests (including a normal coagulation profile), ECGs, vital signs and spirometry.
* Normal spirometry FEV1 (Forced Expiratory Volume in the first second)≥80% of predicted, FEV1/Forced Vital Capacity (FVC) ratio ≥70%) at screening
* Non-smokers for at least one year and with a smoking history of less than 5 pack-years [number of pack years = (number of cigarettes per day/20) x number of years smoked].
* Body weight of ≥50 kg and a body mass index BMI (body mass index) of 20 to 24.9 kg/m2
* Height 170 to 195 cm

Exclusion Criteria:

* Significant history of or current cardiovascular, respiratory (eg asthma, chronic obstructive pulmonary disorder (COPD), bronchiectasis, active Tuberculosis [TB]), hepatic, renal, gastrointestinal, endocrine, hematological, autoimmune or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* Skin lesions in the area used for the dermal application such as dermographism, dermatitis or eczema.
* Use of prescription or non-prescription drugs (except paracetamol), including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days or 5 half-lives (whichever is longer) before the first dose of study medication, unless, in the opinion of the investigator, the medication will not interfere with the study procedures or compromise participant safety.
* History of sensitivity to enrofloxacin, ciprofloxacin or any other fluoroquinolones, or a history of drug or other allergy that, in the opinion of the investigator, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 3 months.
* The participant has participated in a clinical trial and has received an investigational product within the following time period before the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Regular use of known drugs of abuse or a positive drugs of abuse test at screening, positive cotinine test at screening
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Upper or lower respiratory tract infection 4 weeks prior to screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
maximum concentration of enrofloxacin in plasma | change of maximum plasma concentration of enrofloxacin baseline to post dose: 5 minutes (m), 10m, 15m, 20m, 30m, 45m, 1 hour (h) , 1,5 h, 2 h, 3h, 4h, 6h, 8h, 12 h, 24 h.
  maximum concentration of enrofloxacin in plasma
Pharmacokinetic assessment of enrofloxacin in urine | change of maximum plasma concentration of enrofloxacin baseline to post dose in urine collection samples : 0-4 hours (h) post, 8-12 hours post, 12-24 hours post
  maximum concentration of enrofloxacin in Urine

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Badorrek, MD, Principal Investigator — Fraunhofer ITEM
Locations (1):
- Fraunhofer Institute for Toxicology and Experimental Medicine, Hanover, Germany